CLINICAL TRIAL: NCT05053841
Title: Implication of Combined Adjuvant Metformin and Aromatase Inhibitor in Overweight or Obese Postmenopausal Breast Cancer Women
Brief Title: Implication of Metformin Plus Aromatase Inhibitor in Obese Postmenopausal Breast Cancer Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Aya Ahmed El Attar, Dr Aya Ahmed El Attar, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22014
Record Dates: First submitted 2021-09-13; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-08

CONDITIONS: Metformin; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Metformin

ARMS (3):
- Control group (No Intervention): fifteen obese females who received letrozole only
- metformin group (Active Comparator): fifteen obese females who received the same dose of letrozole plus metformin (2000 ± 500) mg daily
  Interventions: Drug: Metformin
- lean group (No Intervention): fifteen non- obese breast cancer females who received letozole for six months, treatment period

INTERVENTIONS:
Drug: Metformin
  Other Names: Glucophage
  Arms: metformin group

SUMMARY:
Metformin is an anti-diabetic oral hypoglycemic agent that considered the gold standard therapy for the treatment of type 2 diabetes. Retrospective analyses show that metformin can offer therapeutic benefits to patients with several forms of cancer. It also has positive weight reducing effect on non-diabetic patient by improving insulin sensitivity (although the exact underlying pathomechanisms remain to be elucidated).

DETAILED DESCRIPTION:
This prospective controlled study aimed to evaluate the effect of combined metformin adjuvant therapy and aromatase inhibitors (letrozole) in postmenopausal obese breast cancer women. In addition, to evaluate the effect of weight reduction on aromatase inhibitor efficacy.

Patients and methods: From February 2014 to June 2015, 75 Post-menopausal breast cancer females' patients were recruited, 53 patients underwent randomization and 45 patients completed six months, treatment. Aromatase inhibitor (letrozole) was administered as once daily in accordance to one of the three groups. Control group: fifteen obese females who received letrozole only; metformin group: fifteen obese females who received the same dose of letrozole plus metformin (2000 ± 500) mg daily, and lean group: fifteen non- obese breast cancer females who received letozole for six months, treatment period. Blood samples were collected at baseline and after six months of aromatase inhibitors treatment for analysis of serum estradiol, osteocalcin, insulin, leptin, lactate and glucose.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women, postmenopausal is defined either by:

A. Age ≥ 55 years and one year or more of amenorrhea. B. Age < 55 years and one year or more of amenorrhea, with an estradiol assay < 20 pg/ml.

• Patients with breast cancer indicated for hormonal treatment with aromatase inhibitors (overweight 30 > BMI ≥ 25, obese BMI ≥ 30 kg/m2 and non obese BMI between 18 and 25 kg/m2).

Exclusion Criteria:

* • Diabetic patients.

  * Patients with metabolic syndrome.
  * Patients with last menstrual cycle less than one year ago.
  * Patient with conditions predispose to acidosis (heart failure, renal failure).
  * Ovarian radiation treatment with luteinizing hormone-releasing hormone (LH-RH) agonist (goserelin acetate or leuprolide acetate) is not permitted for induction of ovarian suppression.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
change in serum level of the study biomarkers after treatment when compared with baseline values | six months
  measuring the serum levels of the studied biomarkers

REFERENCES:
- [Derived] El-Attar AA, Ibrahim OM, Alhassanin SA, Essa ES, Mostafa TM. Effect of metformin as an adjuvant therapy to letrozole on estradiol and other biomarkers involved in the pathogenesis of breast cancer in overweight and obese postmenopausal women: a pilot study. Eur J Clin Pharmacol. 2023 Feb;79(2):299-309. doi: 10.1007/s00228-022-03444-6. Epub 2022 Dec 23. PMID 36562831